CLINICAL TRIAL: NCT06080906
Title: Immunogenicity and Safety of the Inactivated Rotavirus Vaccine (Vero Cells) in Toddlers and Infants Aged From 2 to 71 Months: A Randomized, Double-blinded, Placebo-controlled Phase II Clinical Trial
Brief Title: Phase II Clinical Trial of the Inactivated Rotavirus Vaccine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Medical Biology, Chinese Academy of Medical Sciences (Other)
Collaborators: Henan Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RV-201
Record Dates: First submitted 2023-10-08; First posted 2023-10-12 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Rotavirus Infections; Diarrhea
Keywords: Rotavirus Infections; Inactivated Rotavirus Vaccine; Diarrhea
MeSH Terms: conditions — Rotavirus Infections; Diarrhea | interventions — Appointments and Schedules

STUDY DESIGN:
Intervention Model Description: 300 toddlers (aged 7-71 months) and 300 infants (aged 2-6 months) will be eligible for parallel enrollment
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tolldlers (7-71 months old, two-dose) (Experimental): Inactivated Rotavirus vaccine (Vero cell) in toddlers aged 7-71 months old on Day 0, 28
  Interventions: Biological: IRV on a 0- and 28-day schedule
- Infants (2-6 months old, three-dose) (Experimental): Inactivated Rotavirus vaccine (Vero cell) in infants aged 2-6 months old on Day 0, 28, 56
  Interventions: Biological: IRV on a 0-, 28- and 56-day schedule
- Placebo in Tolldlers (7-71 months old, two-dose) (Placebo Comparator): Two doses of placebo at the vaccination schedule of Day 0, 28
  Interventions: Biological: Placebo on Day 0, 28
- Placebo in Infants (2-6 months old, three-dose) (Placebo Comparator): Three doses of placebo at the vaccination schedule of Day 0, 28, 56
  Interventions: Biological: Placebo on Day 0, 28, 56

INTERVENTIONS:
Biological: IRV on a 0- and 28-day schedule — Inactivated Rotavirus vaccine (Vero Cells) of 320EU/0.5ml on Day 0, 28
  Arms: Tolldlers (7-71 months old, two-dose)
Biological: IRV on a 0-, 28- and 56-day schedule — Inactivated Rotavirus vaccine (Vero cell) of 320EU/0.5ml on Day 0, 28, 56
  Arms: Infants (2-6 months old, three-dose)
Biological: Placebo on Day 0, 28 — Two doses of placebo at the vaccination schedule of Day 0, 28
  Arms: Placebo in Tolldlers (7-71 months old, two-dose)
Biological: Placebo on Day 0, 28, 56 — Three doses of placebo at the vaccination schedule of Day 0, 28, 56
  Arms: Placebo in Infants (2-6 months old, three-dose)

SUMMARY:
This study is a randomized, double-blinded, placebo-controlled phase 2 clinical trial to evaluate the immunogenicity and safety of Inactivated Rotavirus Vaccine (IRV) in children (aged 2-71 months). Primary immunogenicity endpoints in two age groups are the anti-RV neutralizing antibody geometric mean titers (GMTs) 28 days after the final dose, anti-RV neutralizing antibody geometric mean increase (GMI), and seroconversion rates between baseline and 28 days after the final dose. The secondary safety endpoints are the number of adverse events/reactions within 30 minutes after each dose, the number of solicited adverse events/reactions within 7 days after each dose, the number of unsolicited adverse events/reactions within 28/30 days after each dose, and the number of serious adverse events (SAE) between the first dose up to 6 months after the final dose. The exploratory endpoints are the anti-RV IgG and IgA antibody GMT 28 days after the final dose, GMI and seroconversion rates of anti-RV IgG and IgA antibody between baseline and 28 days after the final dose, GMT and seropositive rates of anti-RV neutralizing antibody, IgG antibody and IgA antibody 90, 180, and 360 days after the final dose. Besides, as the exploratory endpoint, the GMT, GMI, and seroconversion rates of cross-neutralizing antibodies against G3 and G9 type of RV, gene transcription differences in peripheral blood mononuclear cells on Day 0 and 28 after the final dose will be assessed.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, placebo-controlled phase 2 clinical trial to evaluate immunogenicity and safety of IRV performed in 600 subjects (aged 2-71 months). Then, 300 toddlers (aged 7-71 months) and 300 infants (aged 2-6 months) will be eligible for parallel enrollment after assessing through medical history and physical examination. Subjects from each age group will be randomly assigned to the vaccine group or placebo group in a ratio of 3:1, that is, 225 subjects of all age groups will be injected with the vaccine while 75 subjects with the placebo.

Toddlers (aged 7-71 months) will receive an injection of the vaccine or placebo in the anterolateral midthigh or deltoid muscle of the upper arm on Day 0 and 28. Infants (aged 2-6 months) will receive an injection of the vaccine or placebo in the anterolateral midthigh or deltoid muscle of the upper arm on Day 0, 28, and 56. There would be 140 subjects in each age group chosen voluntarily for the immune persistence cohort according to the order of enrollment. The duration of toddlers (aged 7-71 months) for intervention is approximately 1 month. Thus, the duration of each subject enrolled in the immune persistence cohort will be approximately 13 months while the duration of the rest of the subjects in the study will be approximately 7 months. The duration of infants (aged 2-6 months) for intervention is approximately 2 months. Thus, the duration of each subject enrolled in the immune persistence cohort will be approximately 14 months while the duration of the rest of the subjects in the study will be approximately 8 months.

For safety assessment, the observation and evaluation of adverse events (AE) from Day 0 to Days 28/30 after each dose, and serious adverse events (SAE) between the first dose up to 6 months after the final dose will be evaluated by diary/contact cards, active reports by subjects' legal guardians, or investigators' phone calls as well as face-to-face visits. Meanwhile, subjects will be observed at the site for at least 30 minutes after each dose. For immunogenicity assessment, neutralizing antibodies against the strain from which the vaccine is based (homologous ZTR-68 strain (G1P[8]), IgG antibodies, IgA antibodies of all subjects, and neutralizing antibodies against the G3 and G9 type RV in 140 subjects of each age group will be assessed. For the exploratory endpoint, the gene transcription level of PBMC will be examined for the preliminary exploration of the possible mechanism of the Inactivated Rotavirus Vaccine (Vero Cells).

ELIGIBILITY:
Inclusion Criteria:

* Age Requirement: Infants and toddlers aged 2 to 71 months at the time of enrollment.
* Provision of Legal Identification: Volunteers and their legal guardians or appointed representatives must provide valid legal identification documents.
* Informed Consent: Legal guardians or appointed representatives of volunteers must have the capacity to understand the informed consent document and the research process, voluntarily participate, sign the informed consent form, and be able to comply with the requirements in the study as well as complete relevant visits on time.
* No Previous Rotavirus Vaccination: Infants and toddlers enrolled in the study should not have received any rotavirus vaccines before enrollment.

Exclusion Criteria:

1. First Dose Exclusion Criteria

   Subjects meeting any of the following exclusion criteria will be not eligible for enrollment:
   * Temperature Requirement: Axillary body temperature prior to vaccination is up to 37.3°C or more.
   * Allergic History: Subjects have a history of allergies to any component of the investigational vaccine (e.g., aluminum hydroxide), any history of vaccine allergies, suspected allergies, or any other severe adverse reactions.
   * Vaccine History: Subjects received any inactivated vaccines or subunit vaccines within 7 days (including the 7th day) prior to vaccination with the investigational vaccine, or any other live attenuated vaccines or COVID-19 vaccines within 14 days (including the 14th day) prior to vaccination.
   * Health Conditions: Subjects have known congenital abnormalities, developmental disorders, genetic defects, or severe malnutrition, among other conditions.
   * Immune-Related Diseases: Subjects have compromised primary or secondary immune function, human immunodeficiency virus (HIV) infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), juvenile rheumatoid arthritis (JRA), inflammatory bowel disease, or other autoimmune diseases.
   * Gastrointestinal Conditions: Subjects have a history of intussusception or chronic gastrointestinal diseases.
   * Neurological and Mental Health: Subjects have a history of seizures, convulsions, cerebral palsy, epilepsy, mental illness, or a family history of such conditions.
   * Acute Illness: Subjects have experienced acute illnesses (e.g., fever) within 3 days prior to vaccination with the investigational vaccine.
   * Immune Therapy: Subjects have received immune-enhancing or immune-suppressing therapy within the last 3 months (continuous oral or intravenous administration for more than 14 days) prior to vaccination.
   * Coagulation Abnormalities: Subjects have a history of coagulation disorders (e.g., coagulation factor deficiency, coagulation disorders).
   * Organ Removal History: Subjects have a history of organ removal (e.g., thyroid, pancreas, liver, spleen) or have asplenia syndrome.
   * Participation in Other Clinical Studies: Subjects are currently or have plans to participate in other clinical studies before enrollment.
   * Special Conditions for Children Aged 24 Months and Below: For such children, additional exclusion criteria include difficult birth, resuscitation after suffocation, a history of neurological damage, premature birth (delivery before the 37th week of gestation), and low birth weight (less than 2500 grams).
   * Investigator's Discretion: The final exclusion criterion is the investigator's discretion to determine whether a subject is suitable for participation in the study.
2. Contraindication of the second and third doses of vaccine

   * Severe Adverse Reactions: Subjects experienced severe adverse reactions after receiving the previous vaccine dose.
   * No Longer Meeting Inclusion Criteria or Meeting First Dose Exclusion Criteria: New conditions that disqualify them from meeting inclusion criteria or that meet the exclusion criteria for the first dose occur after receiving the previous dose, as determined by the investigator.
   * Vaccination with Other Rotavirus Vaccines During the Study: Subjects received other rotavirus vaccines during the study period.
   * Other Exclusion Reasons as Determined by the Investigator: The investigator determines other reasons for exclusion.

Ages: 2 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2025-02-17 (Estimated); Study Completion 2025-06-17 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity index-geometric mean titer (GMT) of neutralizing antibody | Day 28 after the second vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method.
Immunogenicity index-geometric mean titer (GMT) of neutralizing antibody | Day 28 after the third vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method.
Immunogenicity index-geometric mean increase (GMI) of neutralizing antibody | Between baseline and day 28 after the second vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method.
Immunogenicity index-geometric mean increase (GMI) of neutralizing antibody | Between baseline and day 28 after the third vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method.
Immunogenicity index-seroconversion rates of neutralizing antibody | Between baseline and day 28 after the second vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method. Seroconversion will be defined as a change from seronegative (<1:8) to seropositive (≥1:8), or a ≥4-fold increase from baseline.
Immunogenicity index-seroconversion rates of neutralizing antibody | Between baseline and day 28 after the third vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method. Seroconversion will be defined as a change from seronegative (<1:8) to seropositive (≥1:8), or a ≥4-fold increase from baseline.

SECONDARY OUTCOMES:
Safety index-incidence of adverse reactions/events | 0-30 minutes after the first dose vaccination
  Incidence of adverse reactions/events after the first dose vaccination.
Safety index-incidence of adverse reactions/events | 0-30 minutes after the second dose vaccination
  Incidence of adverse reactions/events after the second dose vaccination.
Safety index-incidence of adverse reactions/events | 0-30 minutes after the third dose vaccination
  Incidence of adverse reactions/events after the third dose vaccination.
Safety index-incidence of solicited adverse reactions/events | Day 0 to 7 after the first dose vaccination
  Incidence of solicited adverse reactions/events after the first dose vaccination.
Safety index-incidence of solicited adverse reactions/events | Day 0 to 7 after the second dose vaccination
  Incidence of solicited adverse reactions/events after the second dose vaccination.
Safety index-incidence of solicited adverse reactions/events | Day 0 to 7 after the third dose vaccination
  Incidence of solicited adverse reactions/events after the third dose vaccination.
Safety index-incidence of unsolicited adverse reactions/events | Day 0 to 28 after the first dose vaccination
  Incidence of unsolicited adverse reactions/events after the first dose vaccination.
Safety index-incidence of unsolicited adverse reactions/events | Day 0 to 28/30 after the second dose vaccination
  Incidence of unsolicited adverse reactions/events after the second dose vaccination.
Safety index-incidence of unsolicited adverse reactions/events | Day 0 to 30 after the third dose vaccination
  Incidence of unsolicited adverse reactions/events after the third dose vaccination.
Safety index-incidence of serious adverse events | From the beginning of the vaccination up to 6 months after the last vaccination completed
  Occurrence of serious adverse reactions/events after vaccination.

OTHER OUTCOMES:
Immunogenicity index-geometric mean titer (GMT) of IgG antibody | Day 28 after the second vaccination
  IgG antibody assay will be performed using the ELISA method.
Immunogenicity index-geometric mean titer (GMT) of IgG antibody | Day 28 after the third vaccination
  IgG antibody assay will be performed using the ELISA method.
Immunogenicity index-geometric mean increase (GMI) of IgG antibody | Between baseline and day 28 after the second vaccination
  IgG antibody assay will be performed using the ELISA method.
Immunogenicity index-geometric mean increase (GMI) of IgG antibody | Between baseline and day 28 after the third vaccination
  IgG antibody assay will be performed using the ELISA method.
Immunogenicity index-seroconversion rates of IgG antibody | Between baseline and day 28 after the second vaccination
  IgG antibody assay will be performed using the ELISA method. Seroconversion will be defined as a change from seronegative (≤1:16) to seropositive (>1:16), or a ≥4-fold increase from baseline.
Immunogenicity index-seroconversion rates of IgG antibody | Between baseline and day 28 after the third vaccination
  IgG antibody assay will be performed using the ELISA method. Seroconversion will be defined as a change from seronegative (≤1:16) to seropositive (>1:16), or a ≥4-fold increase from baseline.
Immunogenicity index-geometric mean titer (GMT) of IgA antibody | Day 28 after the second vaccination
  IgA antibody assay will be performed using the ELISA method.
Immunogenicity index-geometric mean titer (GMT) of IgA antibody | Day 28 after the third vaccination
  IgA antibody assay will be performed using the ELISA method.
Immunogenicity index-geometric mean increase (GMI) of IgA antibody | Between baseline and day 28 after the second vaccination
  IgA antibody assay will be performed using the ELISA method.
Immunogenicity index-geometric mean increase (GMI) of IgA antibody | Between baseline and day 28 after the third vaccination
  IgA antibody assay will be performed using the ELISA method
Immunogenicity index-seroconversion rates of IgA antibody | Between baseline and day 28 after the second vaccination
  IgA antibody assay will be performed using the ELISA method. Seroconversion will be defined as a change from seronegative (<1:8) to seropositive (≥1:8), or a ≥4-fold increase from baseline.
Immunogenicity index-seroconversion rates of IgA antibody | Between baseline and day 28 after the third vaccination
  IgA antibody assay will be performed using the ELISA method. Seroconversion will be defined as a change from seronegative (<1:8) to seropositive (≥1:8), or a ≥4-fold increase from baseline.
Immunogenicity index-geometric mean titer (GMT) of IgG antibody | Day 90,180 and 360 after the second vaccination
  IgG antibody assay will be performed using the ELISA method.
Immunogenicity index-geometric mean titer (GMT) of IgG antibody | Day 90,180 and 360 after the third vaccination
  IgG antibody assay will be performed using the ELISA method.
Immunogenicity index-seropositive rates of IgG antibody | Day 90,180 and 360 after the second vaccination
  IgG antibody assay will be performed using the ELISA method. Seropositivity will be defined as the seropositive results (>1:16).
Immunogenicity index-seropositive rates of IgG antibody | Day 90,180 and 360 after the third vaccination
  IgG antibody assay will be performed using the ELISA method. Seropositivity will be defined as the seropositive results (>1:16).
Immunogenicity index-geometric mean titer (GMT) of IgA antibody | Day 90,180 and 360 after the second vaccination
  IgA antibody assay will be performed using the ELISA method.
Immunogenicity index-geometric mean titer (GMT) of IgA antibody | Day 90,180 and 360 after the third vaccination
  IgA antibody assay will be performed using the ELISA method.
Immunogenicity index-seropositve rates of IgA antibody | Day 90,180 and 360 after the second vaccination
  IgA antibody assay will be performed using the ELISA method. Seropositivity will be defined as the seropositive results (≥1:8).
Immunogenicity index-seropositive rates of IgA antibody | Day 90,180 and 360 after the third vaccination
  IgA antibody assay will be performed using the ELISA method. Seropositivity will be defined as the seropositive results (≥1:8).
Immunogenicity index-geometric mean titer (GMT) of neutralizing antibody | Day 90,180 and 360 after the second vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method.
Immunogenicity index-geometric mean titer (GMT) of neutralizing antibody | Day 90,180 and 360 after the third vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method.
Immunogenicity index-seropositive rates of neutralizing antibody | Day 90,180 and 360 after the second vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method. Seropositivity will be defined as the seropositive results (≥1:8).
Immunogenicity index-seroconversion rates of neutralizing antibody | Day 90,180 and 360 after the third vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method. Seropositivity will be defined as the seropositive results (≥1:8).
Immunogenicity index-geometric mean titer (GMT) of cross- neutralizing antibody | Day 28 after the second vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method.
Immunogenicity index-geometric mean titer (GMT) of cross-neutralizing antibody | Day 28 after the third vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method.
Immunogenicity index-geometric mean increase (GMI) of cross-neutralizing antibody | Between baseline and day 28 after the second vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method.
Immunogenicity index-geometric mean increase (GMI) of cross-neutralizing antibody | Between baseline and day 28 after the thrid vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method.
Immunogenicity index-seroconversion rates of cross-neutralizing antibody | Between baseline and day 28 after the second vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method. Seroconversion will be defined as a change from seronegative (<1:8) to seropositive (≥1:8), or a ≥4-fold increase from baseline.
Immunogenicity index-seroconversion rates of cross-neutralizing antibody | Between baseline and day 28 after the thrid vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method. Seroconversion will be defined as a change from seronegative (<1:8) to seropositive (≥1:8), or a ≥4-fold increase from baseline.
mRNA sequencing analysis of peripheral blood monouclear cells（PBMCs） | Between baseline and day 28 after the third vaccination
  Differentially expressed genes of infants（2-6 months）between baseline and day 28 after the third vaccination will be measured by mRNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Yanxia Wang, Principal Investigator — Henan Center for Disease Control and Prevention
Locations (1):
- Tongxu Center for Disease Prevention and Control, Kaifeng, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided